CLINICAL TRIAL: NCT04171843
Title: A Phase 1/2a, Open-label, Dose-escalation, Dose-expansion Study to Evaluate the Safety and Clinical Activity of PBCAR269A, With or Without Nirogacestat, in Study Participants With Relapsed/Refractory Multiple Myeloma
Brief Title: A Dose-escalation Study to Evaluate the Safety and Clinical Activity of PBCAR269A, With or Without Nirogacestat, in Study Participants With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to lack of sufficient therapeutic effect
Sponsor: Precision BioSciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PBCAR269A-01
Record Dates: First submitted 2019-11-12; First posted 2019-11-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine; Cyclophosphamide; nirogacestat

STUDY DESIGN:
Intervention Model Description: In Phase I, 3 escalating dose groups will be enrolled and treated sequentially, with the possibility of a single de-escalation. Within each dose group, at least 3 and at most 6 study participants will be treated with a single dose of PBCAR269A using a standard 3 + 3 design. The starting dose of PBCAR269A will be 6 x 105 CAR T cells/kg body weight. Subsequent dose groups will be treated with escalating doses to a maximum dose of 6 x 106 CAR T cells/kg. In the absence of DLTs, the dose will be increased using a fixed-dose scheme.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- PBCAR269A at Dose Level 1 (Cohort A) (Experimental): The starting dose of PBCAR269A will be 6 x 10^5 CAR T cells/kg body weight.
  Interventions: Genetic: PBCAR269A; Drug: Fludarabine; Drug: Cyclophosphamide
- PBCAR269A at Dose Level 2 (Experimental): 2 × 10^6 CAR T cells/kg body weight.
  Interventions: Genetic: PBCAR269A; Drug: Fludarabine; Drug: Cyclophosphamide
- PBCAR269A at Dose Level 3 (Experimental): 6 × 10^6 CAR T cells/kg body weight.
  Interventions: Genetic: PBCAR269A; Drug: Fludarabine; Drug: Cyclophosphamide
- PBCAR269A at Dose Level 2 (Cohort B) (Experimental): 2 × 10^6 CAR T cells/kg body weight.
  Interventions: Genetic: PBCAR269A; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Nirogacestat
- PBCAR269A at Dose Level 1 (Cohort B) (Experimental): 6 x 10^5 CAR T cells/kg body weight.
  Interventions: Genetic: PBCAR269A; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Nirogacestat
- PBCAR269A at Dose Level 3 (Cohort B) (Experimental): 6 × 10^6 CAR T cells/kg body weight.
  Interventions: Genetic: PBCAR269A; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Nirogacestat

INTERVENTIONS:
Genetic: PBCAR269A — Allogeneic anti-BCMA CAR T-cell
Drug: Fludarabine — Fludarabine is used for lymphodepletion.
Drug: Cyclophosphamide — Cyclophosphamide is used for lymphodepletion.
Drug: Nirogacestat — Allogeneic anti-BCMA CAR T-cell
  Arms: PBCAR269A at Dose Level 1 (Cohort B); PBCAR269A at Dose Level 2 (Cohort B); PBCAR269A at Dose Level 3 (Cohort B)

SUMMARY:
This is a Phase 1/2a, nonrandomized, open-label, parallel assignment, single-dose, dose-escalation, and dose-expansion study to evaluate the safety and clinical activity of PBCAR269A, with or without nirogacestat, in adults with r/r MM. Study subjects in Cohort A will receive PBCAR269A and study subjects in Cohort B will receive PBCAR269A and nirogacestat. At each dose level, study subjects in Cohort A and Cohort B will receive the same dose of PBCAR269A. In Cohort B, all study subjects will follow the same dosing regimen of nirogacestat. This study was terminated prior to beginning of Phase II due to lack of sufficient therapeutic effect

DETAILED DESCRIPTION:
This is a multicenter, nonrandomized, open-label, parallel assignment, single-dose, dose-escalation, and dose-expansion study to evaluate the safety and clinical activity of PBCAR269A, with or without nirogacestat, in adults with r/r MM. Before initiating the study treatment PBCAR269A, all study participants will be administered lymphodepletion chemotherapy. The initial lymphodepletion chemotherapy regimen will be composed of fludarabine and cyclophosphamide during the Screening Period. Study subjects in Cohort B will also receive nirogacestat. On Day 0 of the Treatment Period, study participants will receive a single intravenous (IV) infusion of PBCAR269A. All subjects are monitored during the treatment period through Day 28. All subjects who receive a dose of PBCAR269A, with or without nirogacestat, will be followed in a separate long-term follow-up (LTFU) study for 15 years after exiting this study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MM with relapsed and/or refractory disease according to the IMWG criteria.
2. Measurable disease at Screening including at least 1 of the criteria below. Note: Study participants with immunoglobulin (Ig) A myeloma in whom serum protein electrophoresis is deemed unreliable due to comigration of normal serum proteins with the paraprotein in the beta region may be considered eligible provided total serum IgA level is >400 mg/dL.

   1. Serum myeloma (M)-protein ≥0.5 g/dL or, urine M-protein >200 mg/24 hour.
   2. Serum free light chain >10mg/dL with abnormal kappa:lambda ratio.
   3. Imaging consistent plasmacytoma and the presence of any clonal plasma cells in peripheral blood or bone marrow.
3. Study participants must be refractory to 2 prior MM treatment regimens including an immunomodulatory imide drug and a protease inhibitor prior to entering the study. Study participants must have recovered or stabilized to Grade ≤2 from any AEs experienced during prior treatment with the exception of neuropathy. Prior therapy requirements are as follows:

   1. Undergone ≥1 complete cycle of treatment for each regimen, unless progressive disease was the best response to the regimen.
   2. Must have received an immunomodulatory agent, a proteasome inhibitor, and an anti- CD38 antibody.
   3. Study participants who are not candidates for ≥1 of the above treatments may still be considered eligible.
4. Has an Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
5. Has adequate bone marrow, renal, hepatic, pulmonary, and cardiac function defined as:

   1. Estimated glomerular filtration rate >30 mL/min/1.73 m2. A 24-hour urine collection for creatinine clearance may be used at the investigator's discretion.
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels both

      ≤3 times of upper limit of normal, unless there is suspected disease in the liver, in which case, no limit is set provided serum bilirubin is within eligibility criterion.
   3. Total bilirubin <2.0 mg/dL, except in study participants with Gilbert's syndrome.
   4. Platelet count >50,000/μL (platelet transfusions acceptable); neutrophils >750/μL.
   5. Left ventricular ejection fraction (LVEF) >45% as assessed by echocardiogram (ECHO) or multiple gated acquisition (MUGA) scan performed within 1 month before starting lymphodepleting chemotherapy. ECHO results performed within 6 months before Screening and at least 28 days after the last cancer treatment may be acceptable if the study participant has not received any treatment with cardiotoxicity risks.
   6. No clinically significant evidence of pericardial effusion or pleural effusion based on investigator's opinion.
   7. Baseline oxygen saturation >92% on room air.
   8. Pulmonary function tests including forced expiratory volume at 1 sec, forced vital capacity, total lung capacity, diffusion capacity of lung for carbon monoxide ≥50% of predicted values. Study participant characteristics
6. All study participants must be willing to practice birth control and refrain from donating sperm or oocytes from the time of enrollment in this study through 6 months after receiving the study treatment.
7. Women of childbearing potential (WOCBP) must test negative for pregnancy at Screening because of the potentially harmful effects of the preparative chemotherapy to the fetus. WOCBP are defined as any women who are not postmenopausal or who have not had a hysterectomy. Postmenopausal is defined as women over the age of 55 who have not had a menstrual period for ≥1 year.
8. Capable of giving signed informed consent.

Exclusion Criteria:

1. Study participant has clinically significant organ involvement by amyloid protein.
2. Study participant has plasma cell leukemia, Waldenstrom's macroglobulinemia, or POEMS syndrome.
3. History of class III or IV congestive heart failure or severe non-ischemic cardiomyopathy, unstable or poorly controlled angina, myocardial infarction, or ventricular arrhythmia within the previous 6 months of starting study treatment.
4. History or presence of clinically relevant central nervous system (CNS) pathology.
5. Active uncontrolled fungal, bacterial, viral, protozoal, or other infection.
6. Any form of primary immunodeficiency (e.g., severe combined immunodeficiency disease).
7. History of human immunodeficiency virus (HIV) infection.
8. Active hepatitis B or hepatitis C confirmed by polymerase chain reaction (PCR). Study participant positive for inactive hepatitis B will be allowed to enroll if on prophylactic treatment.
9. History of hypertension crisis or hypertensive encephalopathy within 3 months prior to Screening.
10. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
11. Abnormal findings during the Screening Period or any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might jeopardize the study participant's safety.
12. History of genetic syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman-Diamond syndrome, or any other known bone marrow failure syndrome.
13. Study participants with active hemolytic anemia.
14. Study participant has received autologous stem cell transplant within 12 weeks of Screening or an allogeneic stem cell transplant within 6 months of starting study treatment. Study participants who have received an allogeneic transplant must be off all immunosuppressive medications for 6 weeks without signs of GvHD.
15. Study participants with second malignancies in addition to MM if the second malignancy has required treatment within the last 3 years or is not in complete remission, with the exception of non-metastatic basal cell or squamous cell skin carcinoma.
16. Study participant has received systemic biologic agent within 28 days. Participation in non-interventional registries or epidemiological studies is not excluded.
17. Study participant has received live vaccine within 4 weeks before Screening. Non-live virus vaccines are not excluded.
18. Before initiation of lymphodepletion, study participants must have recovered or stabilized to Grade ≤2 from any AEs experienced during prior treatment with the exception of neuropathy.
19. Radiotherapy within 4 weeks before Screening should be discussed with the monitor.
20. Presence of pleural/peritoneal/pericardial catheter.
21. Current use of any anticoagulant or antiplatelet therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of PBCAR269A | Day 1 - Day 28
  To determine the maximum tolerated dose (MTD), which is defined as the dose level at which fewer than 33% of patients experience a dose limiting toxicity (DLT) using a 3+3 strategy.

SECONDARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity(ies) | 1 year
  To assess adverse events as dose limiting toxicities as defined by the protocol and CTCAE v5.0.
Objective Response Rate of Patients | 1 year
  To assess ORR to treatment with PBCAR269A through Day 360 will be noted using the IMWG response criteria.
  The ORR is defined as the proportion of study participants meeting the definition of response within the study population to the response evaluable population. ORR will be summarized by number and percentage of study participants meeting the definition of ORR along with the corresponding exact 95% CIs. DoR, defined as the duration (days) from initial response to disease relapse, progression, or death will be descriptively analyzed using Kaplan-Meier methods. The number of study participants achieving DoR at 3, 6, 9, and 12 months will also be calculated. Exploratory efficacy analyses include changes from Baseline in CBC counts, CAR T cells, cytokines, and CRP levels.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Vainorius, MD, Study Chair — Precision BioSciences, Inc.
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - University of California San Francisco, San Francisco, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - MD Anderson, Houston, Texas